CLINICAL TRIAL: NCT06074029
Title: Exploratory Study on the Therapeutic Effect Prediction Model of Immune Checkpoint Inhibitors for Advanced Biliary Tract Cancer
Brief Title: Exploratory Study on the Therapeutic Effect Prediction Model of Advanced BTC Immunotherapy
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Geneplus-Beijing Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: JYJ-001
Record Dates: First submitted 2023-09-24; First posted 2023-10-10 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Biliary Tract Cancer; Immune Checkpoint Inhibitor; Predictive Cancer Model
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immunotherapy cohort (Experimental): Patients who were administered with immunotherapy
  Interventions: Drug: Immune Checkpoint Inhibitors

INTERVENTIONS:
Drug: Immune Checkpoint Inhibitors — Immune Checkpoint Inhibitors including Durvalumab, Pembrolizumab and Toripalimab

SUMMARY:
1. Establish a predictive model for the efficacy of immune checkpoint inhibitors (ICI) in Chinese patients with biliary tract cancers. By analyzing the dynamic changes of circulating tumor DNA (ctDNA) and other clinical and pathological features before and after ICI treatment in a cohort of patients with biliary tract tumors, a predictive model can be established to evaluate the efficacy of ICI treatment in the early stages or even before treatment, serving as a reliable tool for selecting patients who are likely to benefit from ICI treatment.
2. Investigate the clinical features of populations that benefit from different immune combination therapies. By comparing the differences and enrichment of mutations between patients receiving different treatment regimens, and if patients have sufficient pre-treatment tissue, further comparisons of differentially expressed genes and pathways may be made.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily participate in the study and agree to sign the informed consent form, are compliant, and cooperate with follow-up.
* Patients with advanced biliary tract cancers (including gallbladder cancer, intrahepatic cholangiocarcinoma (ICC), hilar cholangiocarcinoma, or distal cholangiocarcinoma) with histologically, cytologically, or clinically confirmed.
* Patients who have undergone curative surgery and experienced disease recurrence after more than 6 months; or patients who have completed adjuvant therapy (chemotherapy and/or radiotherapy) and have been disease-free for more than 6 months after completing adjuvant therapy are eligible for inclusion.
* Regardless of gender, age 18-80 years old.
* ECOG PS of 0-2 with expected survival time ≥12 weeks.
* According to RECIST V1.1, the patient had at least one measurable lesion.
* The patient is suitable for treatment with immune checkpoint inhibitors (PD-1/PD-L1 inhibitor).

Exclusion Criteria:

* Suffering from other malignant tumors.
* Previous systemic treatment received.
* Patients with serious organic diseases cannot receive the treatment designed in this study;
* Having a psychiatric disorder does not guarantee compliance with this study.
* Patients with symptomatic brain metastasis or complications related to brain metastasis or cognitive impairment.
* Adverse events (except hair loss of any grade) from previous antitumor therapy did not return to ≤ grade 1 or better (According to CTCAE version 5.0).
* Previously received any cell or organ transplant treatment.
* Allergy to the therapeutic drugs of this study or CT or MRI-enhanced contrast agents.
* Received local hepatobiliary treatment (including various types of ablations, percutaneous ethanol or acetic acid injection, high-intensity focused ultrasound, transarterial embolization, chemotherapy, or chemoembolization) within 14 days before the start of the study treatment.
* The physician determines that there are any contraindications to ICI treatment.
* During the second blood monitoring, the disease changes could not be judged (such as unexplained ascites, worsening symptoms); Or non-disease progression, but the next immunotherapy is not planned.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | Baseline up to approximately 12 months
  It refers to the time from the first administration of the regimen to the first occurrence of disease progression or death due to any cause in the subjects.

SECONDARY OUTCOMES:
Objective response rate | Baseline up to approximately 6 months
  The proportion of patients whose tumor volume shrinks to a predetermined value and can maintain the minimum required duration, including complete response and partial response.
Overall survival | Baseline up to approximately 15 months
  The time from randomization to death due to any cause in the subjects.
Time to treatment discontinuation | Baseline up to approximately 12 months
  The time from the beginning of ICI drug use to the cessation of ICI drug use for any reason

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences & Peking Union Medical College Hospital (CAMS&PUMCH), Beijing, Beijing Municipality, China